CLINICAL TRIAL: NCT07249099
Title: Cohort of Cord Blood Bank (CCBN)
Brief Title: Cohort of Cord Blood Bank
Status: Enrolling by invitation | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: QTJC2025029
Record Dates: First submitted 2025-08-01; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-03

CONDITIONS: Health Status; Childhood Diseases
Keywords: umbilical cord blood; Health status of people stored umbilical cord blood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of this observational study was to establish a cohort of umbilical cord blood stored in Tianjin Cord Blood Bank.

DETAILED DESCRIPTION:
This is an observational study. It is planned to observe the incidence and death of common chronic non-communicable diseases, rare diseases and key diseases through follow-up of environmental exposure in the early life of the study population and investigation of adverse lifestyle of mothers during pregnancy, and explore the influence of factors including genetics, environment and lifestyle on the occurrence, development and prognosis of the diseases concerned.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participated in this study and provided signed informed consent forms.
* People stored umbilical cord blood in Tianjin Cord Blood Bank.
* The information registered at the time of storage is complete and the contact details are genuine and available.

Exclusion Criteria:

* Refusing to answer the researcher's phone or refusing to accept the investigation.
* People who are unable or unsuitable to participate in the study for various other reasons .

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: People stored umbilical cord blood in Tianjin Cord Blood Bank
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Health status | The diseases status of participants will be assessed at baseline and at follow-up visits every 3 to 5 years, up to 10 years. The events include the occurrence of childhood diseases at baseline, as well as disease progression or death during follow-up.
  The health status of people stored umbilical cord blood

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China